CLINICAL TRIAL: NCT02025101
Title: Characterization of Slow Coronary Flow
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0048-13-HYMC
Record Dates: First submitted 2013-12-29; First posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Cardiovascular Abnormalities; Vascular Diseases
Keywords: Slow Coronary Flow
MeSH Terms: conditions — Cardiovascular Abnormalities; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Slow Coronary Flow: Patients who were hospitalized with anginal pain and with laboratory markers or pathological ECG for ischemia.

SUMMARY:
Description of the phenomena "Slow Coronary Flow" (SCF), according to the data that has been collected from patients hospitalized with specific criteria. Clinical follow-up of these patients to determine whether they suffered from any cardial or psychological disorders that might be a result of SCF.

ELIGIBILITY:
Inclusion Criteria:

* anginal pain
* laboratory markers
* pathological ECG for ischemia

Exclusion Criteria:

* obstructed coronary artery during catheterization
* very narrow coronary artery

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were hospitalized with anginal pain
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Collection of characteristics of slow coronary flow from approximately 90 patient records | Six months
  Characteristics of slow coronary flow will be collected from approximately 90 patient medical records and will analyzed to find the common variables. This analysis will show whether there is any statistical significance to these characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Frimerman, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel